CLINICAL TRIAL: NCT03282253
Title: Elevated Stearoyl-CoA Desaturase-1 Expression Predicts the Disease Severity and Clinical Outcomes of Severe Acute Pancreatitis
Brief Title: Elevated Stearoyl-CoA Desaturase-1 Expression Predicts the Disease Severity of Severe Acute Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Weiqin Li, Director of Department of Surgical Intensive Care Unit, Nanjing University School of Medicine
Other Study IDs: ESCDEPDSSAP
Record Dates: First submitted 2017-09-12; First posted 2017-09-13 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Acute Pancreatitis; Organ Failure, Multiple
MeSH Terms: conditions — Pancreatitis; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investgatiors aimed to investigate the associations between serum levels of stearoyl-CoA desaturase-1（SCD-1） and the disease severity as well as the presence of adverse clinical events, such as local complications, organ failure, mortality and so on.In this prospective study, participants were divided into two groups based on serum SCD-1 concentration on admission and prospectively observe the disease severity and clinical outcomes of them.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute pancreatitis (Atlanta standard), abdominal pain occurred within one week of admission;
2. APACHEII score is more than 8 and Ranson score is greater than 3;
3. Age 18-75;
4. Obtaining informed consent.

Exclusion Criteria:

1. Pregnancy pancreatitis;
2. Patients with the following disease history: severe cardiac, pulmonary, renal, liver function insufficiency or immunodeficiency disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with the diagnosis of acute pancreatitis (Atlanta standard), abdominal pain occurred within one week of admission; we intended to include the severer cases (APACHEII score is more than 8 and Ranson score is greater than 3).
Sampling Method: Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
the incidence rate of infected pancreatic necrosis | 2-4 week after disease onset

SECONDARY OUTCOMES:
the incidence rate of organ failure | 1-2 week after disease onset
  the incidence rate of organ failure (transient or persistent)
the incidence rate of local complications | 1-2 week after disease onset
  acute peripancreatic fluid collections, pancreatic pseudocycts, acute necrotic collections and walled-off necrosis